CLINICAL TRIAL: NCT06632730
Title: Therapeutic Management and Current Situation Related to the Use of Resources and Costs of Spinal Muscular Atrophy (SMA) in Spain: A Retrospective, Multicenter Analysis Based on Medical Record Review. TREaSURE Study
Brief Title: Therapeutic Management and Use of Resources and Costs of Spinal Muscular Atrophy in Spain
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: COAV101A1ES05
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Spinal Muscular Atrophy Type I; Spinal Muscular Atrophy Type II
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Spinal Muscular Atrophy (SMA) Cohort: Pediatric patients with SMA type I, SMA type II, or presymptomatic SMA.

SUMMARY:
An observational, retrospective, cross-sectional, multicenter study. Real-world data were obtained from medical records of Spanish public hospitals (9 hospitals).

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with SMA type I or SMA type II.
* Patients with medical records available in the hospital.
* Patients diagnosed with SMA type I or SMA type II after 2017 for whom a minimum of 6 months of follow-up was available.

Exclusion criteria:

• Patients who participated in an experimental design study except for those in the long-term follow-up period, during the observation period.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Cost per Year of Use of Resources for Medical Visits | Up to 12 months
  Medical visits included:
  * Primary care
  * Pediatric neurology
  * Rehabilitation physician
  * Traumatologist
  * Nutritionist
  * Pulmonologist
  * Cardiologist
  * Physical therapist
  * Nursing staff
  * Phoniatrist
  * Speech therapist
  * Rehabilitation sessions
  * Other specialists
  * Total medical visits
  * Hospital emergency room visits
  * Outpatient emergency room visit
  * Hospitalizations/Admissions to ward
  * Hospitalizations due to admissions to the intensive care unit (ICU)
  * Total hospitalizations (ward and ICU)
  * Therapy session separately from medical visits
Costs per Year of Use of Resources for Medical Tests | Up to 12 months
  Medical tests included:
  * Blood count
  * Vitamin D test
  * Blood creatine kinase test
  * Electromyogram
  * Brain magnetic resonance imaging
  * Muscle magnetic resonance imaging
  * Bone densitometry
  * Nocturnal polysomnography
  * Muscle biopsy
  * Nerve conduction velocity study
  * Blood amino acid test
  * DNA test to confirm diagnosis
  * Total additional tests
Cost per Year of Use of Resources for Treatment | Up to 12 months
  Treatments included:
  * Nusinersen (loading and maintenance dose)
  * Total Nusinersen
  * Risdiplam
  * Onasemnogene abeparvovec
  * Total treatments for SMA
  * Palivizumab
  * Influenza vaccine
  * Meningococcal vaccine
  * High protein shakes
  * Total adjuvant treatments
  * Total treatments

SECONDARY OUTCOMES:
Number of Patients per Sociodemographic Category | Baseline
  Sociodemographics included:
  * Biological sex
  * Dead patients
  * Growth percentiles for growth charts (3%, 4-15%, 16-50%, 51-85%, 86-97%, greater than 97%)
  * Patient's cohabitants (father, mother, both parents, brother(s), sister(s), other relatives)
  * Patient's caregiver (father, mother, both parents, brother(s), sister(s), other relatives)
  * Patient's primary caregiver (father, mother, both parents, brother(s), sister(s), other relatives)
Sociodemographic: Age | Baseline
  * Age at the time of data collection
  * Age of onset of SMA symptoms
  * Age at clinical diagnosis of SMA
  * Age of death
Sociodemographic: Weight | Baseline
Sociodemographic: Height | Baseline
Sociodemographic: Body mass index (BMI) | Baseline
Number of Patients per Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * Anti-adeno-associated virus serotype 9 (AAV9) antibody titer test
  * Neonatal screening for SMA together with other screening tests
  * Prenatal or perinatal SMA diagnosis
  * Ventilatory support
  * Patient with scoliosis
  * Patient with scoliosis surgery
  * Patients with a chair for scoliosis
  * Total or partial cost of the chair for scoliosis borne by the family
  * Patients still use a chair for scoliosis at the time of data collection
  * Patients with back brace
  * Total or partial cost of the back brace borne by the family
  * Patient with hip dislocations or subluxations
  * Head control
  * Relevant medical record
  * End of ventilatory support
Clinical Characteristic: Age From Which Information Was Available | Baseline
Clinical Characteristic: Time From Onset of Symptoms to Diagnosis | Baseline
  Time intervals included:
  * Less than 1 month
  * 1 to 3 months
  * 4 to 6 months
  * 7 to 18 months
  * More than 18 months
Clinical Characteristic: Number of Patients Categorized by International Classification of Diseases (ICD) Code | Baseline
  ICD codes included:
  * ICD-9 335.1: Spinal muscular atrophy
  * ICD-9: 335.1: Spinal muscular amyotrophy, unspecified
  * ICD-9 335.11: Kugelberg-Welander disease
  * ICD-10 G12.1: Other hereditary spinal muscular atrophies
  * ICD-10 G12.25: Progressive spinal muscular atrophy
  * ICD-10 G12.8: Other spinal muscular atrophies and related syndromes
  * ICD-10 G12.9: Spinal muscular atrophy, unspecified
Clinical Characteristic: Number of Patients Categorized by Type of Diagnosis of Muscle Atrophy | Baseline
  Diagnosis types included:
  * Clinical suspicion and subsequent patient referral for genetic confirmation
  * Genetic diagnosis
Clinical Characteristic: Number of Patients Categorized by Type of Mutation | Baseline
  Mutations included:
  * Biallelic deletion of exons
  * Biallelic deletion of exon 7
  * Biallelic deletion of exons 7 and 8
  * Compound heterozygous mutation
  * Point mutation and deletion of exons 7 and 8
  * Biallelic point mutation
Clinical Characteristic: Number of Patients Categorized by Survival of Motor Neuron 2 (SMN2) Gene Copy Number | Baseline
  SMN2 copy numbers: 0, 1, 2, 3, 4, and greater than 4.
Clinical Characteristic: Number of Patients Categorized by SMA-associated Comorbidities | Baseline
  SMA-associated comorbidities included:
  * Chronic lung disease
  * Swallowing impairment
  * Malnutrition
  * Hypoxic encephalopathy
  * Relapsing obstructive bronchial syndrome
  * Recurrent pneumonia
  * Sleep apnea-hypopnea syndrome
  * Epilepsy
  * Hip dysplasia
  * Obesity
  * Respiratory compromise
  * Thorax deformity
  * Scoliosis
  * Other
Clinical Characteristic: Number of Patients Categorized by Family History of SMA | Baseline
  Family history categories included:
  * Yes
  * No
  * Mother
  * Father
  * Both parents
  * Brothers and sisters
  * Other
Clinical Characteristic: Number of Patients Categorized by Type of Ventilatory Support | Baseline
  Types of ventilatory support included:
  * Invasive (hospital and outpatient)
  * Non-invasive (hospital and outpatient)
Clinical Characteristic: Number of Patients Categorized by Reason of Ventilatory Support Regimen | Baseline
  Reasons of ventilatory support included:
  * Preventive intent
  * Therapeutic intent
Clinical Characteristic: Duration of Ventilatory Support | Baseline
Clinical Characteristic: Number of Patients With Nutritional Supplementation | Baseline
Clinical Characteristic: Number of Patients Categorized by Type of Administration of Nutritional Supplementation | Baseline
  Types of administration included:
  * By mouth
  * Through a feeding tube
  * Both (mouth and feeding tube)
  * Through gastrostomy
Clinical Characteristic: Number of Patients Categorized by Type of Nutritional Supplementation Received by Mouth | Baseline
  Types of nutritional supplementation included liquid thickeners (corn starch and Nutilis Clear thickener, neutral taste, Nutricia) and nutrition supplements (Resource shakes, High protein shakes, Ensure Junior drink, Infatrini, Pediasure Complete, RESOURCE C, Vitamin D, Fortini high protein shakes, protein shakes, Pediasure, Resource with fiber, Resource protein).
Clinical Characteristic: Number of Patients Who Received Liquid Thickener and Nutritional Supplements by Mouth | Baseline
Clinical Characteristic: Number of Patients Who Received Liquid Thickener and Nutritional Supplements Through a Feeding Tube | Baseline
Clinical Characteristic: Duration of Nutritional Supplementation Received by Mouth and Through a Feeding Tube or Gastrostomy | Baseline
Clinical Characteristic: Number of Surgeries for Patients With Scoliosis | Baseline
Clinical Characteristic: Number of Patients Categorized by Type of Surgery Received for Scoliosis | Baseline
  Types of surgeries included:
  * Growing rods lengthening
  * Dorsal/lumbar dorsal arthrodesis
  * Growing rods
Clinical Characteristic: Number of Patients Categorized by Type of Joint Contracture | Baseline
  Types of joint contractures included proximal and distal.
Clinical Characteristic: Number of Patients Who Reached Each Motor Development Milestone | Baseline
  Developmental Milestones:
  * Sitting independently or with support
  * Standing independently or with support
  * Walking independently or with support
  * Crawling with the elbows, belly crawl, or with hands and knees
Clinical Characteristic: Number of Patients Categorized by Relevant Surgical History in Addition to Scoliosis Surgery Related to SMA Categorized by Type of Surgery | Baseline
  Surgeries included:
  * Mouth surgery
  * Tracheostomy
  * Surgery for gastrostomy
  * Tenotomy
  * Other
Number of Scheduled and Unscheduled Healthcare Visits per Patient per Year | Up to 12 months
  Healthcare visits included:
  * General
  * Primary care
  * Pediatric neurology
  * Rehabilitation physician
  * Traumatologist
  * Nutritionist
  * Pulmonology
  * Cardiologist
  * Physical therapy
  * Nursing staff
  * Phoniatrist
  * Speech therapist
  * Rehabilitation sessions
  * Other experts
  * Emergency Room
  * Related to therapy
Total Number of Scheduled and Unscheduled Healthcare Visits per Patient per Year | Up to 12 months
Number of Scheduled and Unscheduled SMA-related Medical Visits | Up to 12 months
  SMA-related medical visits included:
  * Primary care
  * Pediatric neurology
  * Rehabilitation physician
  * Traumatologist
  * Nutritionist
  * Pulmonologist
  * Cardiologist
  * Physical therapist
  * Nursing staff
  * Phoniatrist
  * Speech therapist
  * Rehabilitation sessions
  * Other specialists
Number of SMA-related Emergency Room Visits | Up to 12 months
  SMA-related emergency room visits included outpatient and hospital visits.
Number of SMA-related Hospitalizations | Up to 12 months
  SMA-related hospitalizations included visits to day hospital, admissions to ward, intensive care unit admissions.
Number of Patients Categorized by Reason for Hospitalization | Up to 12 months
  Hospitalization included admission to ward. Reason for hospitalization included related to treatment and not related to treatment.
Number of Patients Categorized by Reason for Admission to Intensive Care Unit (ICU) | Up to 12 months
  Reason for admission to ICU included related to treatment and not related to treatment.
Number of Patients With a Multidisciplinary Follow-up | Up to 12 months
Number of Patients Categorized by Medical Areas Involved in Follow-up | Up to 12 months
  Medical areas included:
  * Pulmonology
  * Endocrinology/nutrition
  * Physical therapy
  * Rehabilitation
  * Logopedics
  * Thoracic surgery
  * Orthopedics
  * Other
Number of Patients Categorized by Type of Additional Tests Needed | Up to 12 months
  Additional tests included:
  * Blood count
  * Vitamin D test
  * Blood creatine kinase test
  * Electromyogram
  * Brain magnetic resonance imaging
  * Muscle magnetic resonance imaging
  * Bone densitometry
  * Nocturnal polysomnography
  * Muscle biopsy
  * Nerve conduction velocity study
  * Blood amino acid test
  * DNA test to confirm diagnosis
Number of Times Each Additional Test Was Performed | Up to 12 months
  Additional tests included:
  * Blood count
  * Vitamin D
  * Blood creatine kinase
  * Electromyogram
  * Brain magnetic resonance imaging
  * Muscle magnetic resonance imaging
  * Bone densitometry
  * Nocturnal polysomnography
  * Muscle biopsy
  * Nerve conduction velocity study
  * Blood amino acid test
  * DNA test to confirm diagnosis
Total Additional Tests | Up to 12 months
Number of Patients Categorized by Type of Treatment for SMA | Up to 6 years and 4 months
  Treatments included:
  * Nusinersen
  * Risdiplam
  * Onasemnogene abeparvovec
  * Palivizumab
  * Influenza vaccine
  * Meningococcal vaccine
  * High protein shakes
Number of Nusinersen Doses | Up to 6 years and 4 months
  Nusinersen doses included loading and maintenance doses.
Risdiplam Dose | Up to 6 years and 4 months
  Risdiplam dose included starting dose and dose changes.
Palivizumab Dose | Up to 6 years and 4 months
Number of High Protein Shakes per Day | Up to 6 years and 4 months
Number of Months of Taking High Protein Shakes | Up to 6 years and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States